CLINICAL TRIAL: NCT03677635
Title: Is There a Relationship Between Memory for Past Events and Motivation for Future Activities?
Brief Title: The Relationship Between Autobiographical Memory and Motivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 214063
Record Dates: First submitted 2017-02-10; First posted 2018-09-19 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2020-02

CONDITIONS: Psychosis
Keywords: Negative Symptoms; Autobiographical Memory
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Guided autobiographical memory recall to enhance specificity and links to the future.
  Interventions: Behavioral: Guided Autobiographical Memory Recall
- Control (No Intervention): Recall without prompts or psychoeducation video.

INTERVENTIONS:
Behavioral: Guided Autobiographical Memory Recall — Participants are asked to recall positive autobiographical memories with the assistance of prompts to promote specificity, generalisability and links to the future. The participants will also view a 5min psychoeducation video on the subject of memory specificity and motivation.
  Arms: Intervention

SUMMARY:
People with a diagnosis of psychosis often experience low motivation and pleasure when thinking about doing future activities. This leads, quite understandably, to doing fewer activities they used to enjoy and not taking up opportunities to do new activities. One model suggests that this may be partly due to difficulties using memories of previous events to help boost motivation and anticipation before a future activity. Research shows that people with psychosis may recall previous events in less detail. These memories therefore may not be as helpful as they could be for motivation. This study will investigate this by asking people with experience of psychosis and low motivation who are seen by a care team in South London and Maudsley NHS Trust to attend two research sessions. In the first session the participants will be asked to recall memories of events from their lives and the researcher will assess how detailed the memories are and how much the participant refers to the past and future. Alongside this task the participants will also be asked to complete measures of symptoms such as low pleasure and motivation as well as a measure of depression. These will be used to find out if the detail and specificity of the memories are related to these symptoms in people with psychosis. The second half of the study will then investigate whether additional prompts to support positive memory retrieval can increase the specificity of this and subsequently improve mood, motivation and self-belief. Participants will be randomised to one of two groups. The clinical group will be guided through their memory recall using prompts and a control group will be asked to recall positive memories without prompts. If the investigators show that supporting memory recall is beneficial then memories for past events may be an important target for future therapies.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of non-affective psychosis (as determined by medical records).
* Above 18yrs old.
* A score of at least 18 on the Clinical Assessment Interview for Negative Symptoms.
* A sufficient command of the English language to engage with the research materials

Exclusion Criteria:

* Lack of capacity to provide informed consent.
* Primary diagnosis of intellectual disability, head injury, substance misuse or known organic cause of psychosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2020-02-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - South London and Maudsley NHS Trust, London
  - Institute of Psychiatry, Psychology & Neuroscience, KCL, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 31 people with a diagnosis of non-affective psychosis participated between May 2017-Feb 2018.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 21 | 10
Completed | 21 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 21 | 10 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.62 (10.98) | 41.10 (9.09) | 39.55 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 16 | 8 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 21 | 9 | 30
  Unknown or Not Reported | 0 | 0 | 0
Clinical Assessment Interview for Negative Symptoms [Mean (Standard Deviation); unit: units on a scale] — The Clinical Assessment Interview for Negative Symptoms (Kring, Gur, Blanchard, Horan, & Reise, 2013) was used to enable the assessment of both experiential and expressive negative symptoms. This takes the form of an interview schedule which is used alongside observations to complete the assessment (13 items, range: 0-52, higher score indicates greater severity of negative symptoms).
  units on a scale | 24.1 (6.37) | 17.1 (6.82) | 21.73 (7.04)

OUTCOME MEASURES:

1. Primary Outcome: Post-Intervention Motivation Score
Description: A rating on a visual analogue scale assessing motivation to repeat the same activity recalled in the future. The scale is rated from 0-100 and a higher score indicated better outcome.
Time Frame: Immediately after completing the intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 21 | 10
units on a scale | 81.01 (4.15) [69.21 to 85.86] | 72.89 (5.79) [65.12 to 88.38]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; Standardised Effect Size; Standardised Effect Size = 0.32, 95% CI 2-sided [.21 to .86]

2. Secondary Outcome: Post-Intervention Anticipatory Pleasure
Description: A rating on a visual analogue scale assessing how pleasant that activity is anticipated to be if repeated. The scale is rated from 0-100 and a higher score indicated better outcome.
Time Frame: Immediately after completing the intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 21 | 10
units on a scale | 84.35 (3.05) | 86.58 (4.76)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other — Cohen's d was reported; Standardised Effect Size; Mean Difference (Final Values) = -.05, 95% CI 2-sided [-.59 to .48]

ADVERSE EVENTS:
Time Frame: 90 mins
Description: Participants were monitored during their participation in the single testing session, which lasted approximately 90 mins, adverse events were not monitored for any period of time after this.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/10
Other Adverse Events (participants affected / at risk) | 0/21 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/35/NCT03677635/Prot_SAP_000.pdf